CLINICAL TRIAL: NCT04799483
Title: The Gemini Study: Study of the Long-Term Safety and Persistence of Cells Following Cell Transfers or Gene Therapy in Identical Twins Discordant for HIV Infection
Brief Title: Safety and Survival of Genetically Modified White Blood Cells in HIV-infected Twins The Gemini Study
Status: Active, not recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020080; 02-I-0080
Record Dates: First submitted 2021-03-15; First posted 2021-03-16 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: HIV
Keywords: Gene Therapy; HIV; Immunotherapy; Syngeneic Cells; Gemini Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study will consolidate under one umbrella protocol all NIH studies of the safety and survival of gene-modified lymphocytes in HIV-infected twins. The major purposes of the current study are to:

* place subjects from the various identical twin cell transfer/gene therapy studies on a single, more uniform schedule of visits;
* examine the long-term safety of apheresis procedures in non-HIV-infected lymphocyte donor twins;
* examine the long-term safety of lymphocytes in HIV-infected lymphocyte recipient twins.

Identical twins enrolled in NIH protocols 93-I-0110, 94-I-0206, 96-HG-0051, and 97-I-0165 involving the transfer of lymphocytes for the treatment of HIV infection are eligible to continue their research participation under the current protocol, 02-I-0080.

Participants will not undergo any additional research procedures in this study. They will continue to take their antiretroviral therapy and will be followed at least once a year, or more often if medically indicated, with a medical history, physical examination and blood tests for routine studies and to determine the number of lymphocytes in the blood. Recipient twins will also have blood levels of gene-modified lymphocytes checked.

Recipient twins will have some blood stored for RCR (replication competent retrovirus) testing, should it become necessary. A special virus was used to insert genes into the donated lymphocytes and, although the virus was rendered incapable of growing in the body, a theoretical risk exists that the virus could mix with other viruses and possibly begin growing or reproducing. If a participant subsequently develops medical problems, the stored blood samples can be checked for RCR to see if it may be a cause of the problem.

DETAILED DESCRIPTION:
Intramural NIAID sponsored several phase I-II studies of cell transfers during the 1990's, including gene-modified cells, in identical twins discordant for HIV infection. These studies were both novel in the field of alternative treatment strategies for HIV infection and served as early studies in the developing field of clinical gene therapy. The current protocol represents an umbrella protocol in which these early trials have been consolidated for purposes of long-term safety monitoring and long-term follow-up of gene-modified cell persistence. Cell recipients as well as donors enrolled in Intramural NIAID twin gene marking, gene therapy and cell transfer studies have been eligible for study participation. Participants are monitored for safety per a uniform standardized schedule. No gene therapy, cell transfers or other investigational therapeutic interventions occur under the auspices of this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:

Activet participation, in an NIAID/CCMD/NHGRI protocol involving the transfer of unmodified lymphocytes, gene-marked lymphocytes or cells containing potentially therapeutic genes in the treatment of HIV-1 infection (cell donors and recipients were eligible).

Ongoing follow-up with a primary medical care provider who manages the subject's HIV-related and/or other medical conditions.

Agree to comply with study requirements and clinical policies.

Able to provide informed consent.

EXCLUSION CRITERIA:

A history of gross noncompliance with prior NIAID/CCMD protocol requirements that, in the opinion of the Principal Investigator, is likely to seriously compromise the safety or value of an individual's participation in the present protocol.

Refusal to follow Clinical Center policy on partner notification (if HIV-positive).

Refusal to permit research blood specimens to be stored (frozen) for potential future studies, including RCR testing will be excluded (participants who have received gene-modified cells may refuse to have specimens stored for research purposes other than RCR).

Any medical condition that, in the opinion of the Principal Investigator, would make the subject inappropriate for protocol participation (such as anemia or inadequate venous access).

Refusal to allow the NIH research team to exchange pertinent medical information with the subjects primary medical care provider.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who participated in the long-term follow-up phase of previous NIAID/NHGRI intramural research protocols in which unmodified cells, gene marked cells or cells with therapeutic genes were infused.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2001-01-05 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the Long-term safety of gene-modified and unmodified infusion | Annually

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Wright, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Donahue RE, Kessler SW, Bodine D, McDonagh K, Dunbar C, Goodman S, Agricola B, Byrne E, Raffeld M, Moen R, et al. Helper virus induced T cell lymphoma in nonhuman primates after retroviral mediated gene transfer. J Exp Med. 1992 Oct 1;176(4):1125-35. doi: 10.1084/jem.176.4.1125. PMID 1383375
- [Background] Carr A, Cooper DA. Adverse effects of antiretroviral therapy. Lancet. 2000 Oct 21;356(9239):1423-30. doi: 10.1016/S0140-6736(00)02854-3. PMID 11052597
- [Background] Morgan RA. Genetic strategies to inhibit HIV. Mol Med Today. 1999 Oct;5(10):454-8. doi: 10.1016/s1357-4310(99)01542-7. PMID 10498914
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2002-I-0080.html